CLINICAL TRIAL: NCT01321489
Title: A Clinical Phase III, Comparative, Open, Multicenter, Prospectively, to Evaluate a Possible Superiority Expressed by the Faster Onset of Action and the Efficacy and Safety of Sildenafil Citrate 20mg Sublingual Tablet, Compared to Viagra ® 50mg Tablet Coated, in the Treatment of Erectile Dysfunction of Different Etiologies
Brief Title: A Study to Evaluate a Possible Superiority Expressed by the Faster Onset of Action and the Efficacy and Safety of Sildenafil Citrate 20mg Sublingual Tablet in the Treatment of Erectile Dysfunction of Different Etiologies
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Laboratório Teuto Brasileiro S/A (Industry)
Responsible Party: Laboratório Teuto Brasileiro S/A, Industry
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TEU-SIL-05/09
Record Dates: First submitted 2011-03-15; First posted 2011-03-23 (Estimated); Last update posted 2011-03-23 (Estimated); Status verified 2011-03

CONDITIONS: Erectile Dysfunction
Keywords: Phase III; Sildenafil Citrate Tablet Sublingual; Erectile dysfunction
MeSH Terms: conditions — Erectile Dysfunction | interventions — Sildenafil Citrate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sildenafil Citrate 20mg Tablet Sublingual (Experimental): Administer one tablet of Sildenafil Citrate 20 mg sublingually 10 minutes before intercourse. It is recommended that the administration of just one tablet a day. The patient will receive six tablets of the medication.
  Interventions: Drug: Viagra ® 50mg tablet Coated
- Viagra ® 50mg tablet Coated (Active Comparator): Administer one tablet of Viagra ® 50mg tablet Coated orally 1 hour before intercourse. It is recommended that the administration of just one tablet a day. The patient will receive six tablets of the medication.
  Interventions: Drug: Sildenafil Citrate 20mg Tablet Sublingual

INTERVENTIONS:
Drug: Sildenafil Citrate 20mg Tablet Sublingual — Administer one tablet of Sildenafil Citrate 20 mg sublingually 10 minutes before intercourse. It is recommended that the administration of just one tablet a day. The patient will receive six tablets of the medication.
  Arms: Viagra ® 50mg tablet Coated
Drug: Viagra ® 50mg tablet Coated — Administer one tablet of Viagra ® 50mg tablet Coated orally 1 hour before intercourse. It is recommended that the administration of just one tablet a day. The patient will receive six tablets of the medication.
  Arms: Sildenafil Citrate 20mg Tablet Sublingual

SUMMARY:
The purpose of this study is to evaluate the tolerability and safety of Sildenafil Citrate 20mg Sublingual tablet, as well as a possible superiority expressed by the faster onset of action compared to Viagra ® 50mg tablet Coated in erectile dysfunction.

DETAILED DESCRIPTION:
Phase III clinical trial, comparative, open, multicenter, prospectively, with random inflow of 78 patients evaluable male patients with erectile dysfunction with IIEF-5 score in between 13 and 24, corresponding to mild or mild to moderate to evaluate the efficacy and safety as well as a possible superiority expressed by the faster onset of action onset of action of study medication.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years;
* Patients with erectile dysfunction of various etiologies (organic, psychogenic and mixed) for at least 6 months;
* Patients with scores in the IIEF-5 between 13 and 24, which correspond to mild or mild to moderate;
* Relationship stable for at least 6 months;
* Patients should be kept with libido;
* Education at least 4 years;
* Do not use sildenafil, vardenafil, tadalafil, lodenafil, injection therapy or vacuum devices up to 72 hours before the screening visit;
* Functions hepatic, hematological, hormonal and renal within the following benchmarks:
* Creatinine: 0.6 to 1.10 mg / dl;
* Urea: 10 - 50mg/dl;
* TGP: up to 40 U / L;
* TGO: ≤ 34 U / L;
* Prolactin: 2.3 to 11.5 ng / ml Men
* Total Testosterone: 241 to 827 ng/100 ml - Men
* Blood glucose: 70 mg / dl and 99mg/dl.

Exclusion Criteria:

* Patients who have failed treatment with inhibitors of phospho-diesterase inhibitors;
* Patients undergoing radical prostatectomy;
* Patients with hypersensitivity to any component of the formula;
* Presence of genital deformities or other disorders that prevent intercourse;
* Operations prior to penile erectile dysfunction or premature ejaculation penis enlargement;
* Use of other treatments for erectile dysfunction or concomitant treatment with nitrates;
* Myocardial infarction or cerebrovascular accident (CVA) for less than 6 months;
* Heart disease or uncontrolled serious;
* Injury cord injury;
* Multiple sclerosis;
* Retinitis pigmentosa;
* Neoplasms known in business and / or treatment;
* History of severe anaphylactic reactions and disease Steven-Johnson;
* Participation in a clinical study in the 2 months prior to inclusion;
* Patients who are making use of antiretrovirals;
* Any other disease or condition is not matched that in the opinion of the investigator, could lead to increased risk for the patient or who makes it inappropriate for this study;
* Comorbidities such as diabetes mellitus, malignant hypertension, blood pressure (BP), systolic> 170 mmHg, diastolic BP levels> 110 mmHg, blood pressure <80 x 50 mmHg, significant cardiovascular disease, alcohol or drugs, or other disorders important.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2011-09; Primary Completion 2012-01 (Estimated); Study Completion 2012-01 (Estimated)

PRIMARY OUTCOMES:
Evaluate a possible superiority expressed by the faster onset of action. | 35 days
  To evaluate a possible superiority expressed by the faster onset of action of Sildenafil Citrate 20mg Tablet Sublingual compared to Viagra ® 50mg tablet Coated in erectile dysfunction.

SECONDARY OUTCOMES:
Evaluate the efficacy and tolerability of Sildenafil Citrate 20mg Sublingual tablet, compared to Viagra ® 50mg tablet Coated in control of Erectile Dysfunction. | 35 days
  The secondary outcame measure will be to evaluate the efficacy and tolerability of Sildenafil Citrate 20mg Sublingual tablet, compared to Viagra ® 50mg tablet Coated in patients with Erectile Dysfunction.

CONTACTS AND LOCATIONS:
Overall Officials: Eduardo Bertero, Investigator, Principal Investigator — Hospital for State Civil Servants of Sao Paulo
Locations (1):
- Ipiranga Hospital, São Paulo, São Paulo, Brazil